CLINICAL TRIAL: NCT04626076
Title: International Registry of Healthcare Workers Exposed to COVID-19 Patients (UNITY Global)
Status: Completed | Type: Observational
Sponsor: Certara (Industry)
Collaborators: Bill and Melinda Gates Foundation (Other); Parexel (Industry)
Responsible Party: Sponsor
Other Study IDs: CER-HCW-001
Record Dates: First submitted 2020-11-10; First posted 2020-11-12 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: SARS-CoV Infection; Covid19
Keywords: SARS-CoV-2 infection; SARS-CoV-2; COVID-19; Healthcare Workers
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Aga Khan University: Pakistan
  Interventions: Other: Comparative Observational Cohort Study
- African Medical and Research Foundation- Uganda: Uganda
  Interventions: Other: Comparative Observational Cohort Study
- African Medical and Research Foundation- Kenya: Kenya
  Interventions: Other: Comparative Observational Cohort Study
- African Medical and Research Foundation- Zambia: Zambia
  Interventions: Other: Comparative Observational Cohort Study
- African Medical and Research Foundation- Senegal: Senegal
  Interventions: Other: Comparative Observational Cohort Study
- 54Gene: Nigeria
  Interventions: Other: Comparative Observational Cohort Study
- African Institute of Biomedical Science & Technology: Zimbabwe
  Interventions: Other: Comparative Observational Cohort Study

INTERVENTIONS:
Other: Comparative Observational Cohort Study — This is a comparative observational cohort study; therefore, no preventive interventions, visits or laboratory tests are mandated. Dosing and duration of potential prophylactic treatment is at the discretion of the institution and/or healthcare provider, in accordance with regular local practice. However, serology testing for SARS-CoV-2 antibodies will be offered to the first 50% of participating HCWs per country, at enrollment and at the last follow-up (i.e. at Week 12)

SUMMARY:
The International Registry of Healthcare Workers Exposed to COVID-19 Patients (UNITY Global), is an international registry of approximately 10,000 healthcare workers in low- and middle-income countries experiencing increasing numbers of COVID-19 cases and commensurate increased exposure to the SARS-CoV-2 virus among their healthcare worker populations.

DETAILED DESCRIPTION:
The registry will enrol HCWs who are experiencing or are expected to experience ongoing and recurrent close contact with confirmed or clinically diagnosed COVID-19 patients. Recruitment for the registry will aim to enrol a representative distribution of HCWs on the front lines of diagnosing and caring for COVID-19 patients in both hospitals and community settings, as well as a balanced sample of HCWs receiving the most commonly administered putatively prophylactic drug regimens.

The registry will collect information on a weekly basis from HCWs across a 12-week period following their first known exposure to confirmed or clinically diagnosed COVID-19 patients prior to or within 30 days after enrollment. Data collection will include the drug regimens being taken by the HCWs, information about their level of exposure to COVID-19 patients, their personal health status, and other factors such as the use of PPE which would likely impact their risk of developing a SARS-CoV-2 infection.

A standard pharmaco-epidemiological inferential analysis will be conducted treating the registry data as a cohort with dynamic exposure to both prophylactic treatment and to COVID-19 infected patients and adjusting for potential confounding. Crude and adjusted hazards ratios will be estimated for each of the prophylactic regimens of interest and any observed impact on the risk of infection among HCWs based on all statistical inferential models will be reported

ELIGIBILITY:
Inclusion Criteria:

Healthcare workers will be entered into this study only if they meet ALL the following criteria:

* Healthcare workers aged ≥ 18 years.
* Healthcare workers must be exposed through ongoing and recurrent contact to a confirmed or clinically diagnosed COVID-19 patient prior to enrollment, or anticipated within 30 days after enrollment.
* Healthcare workers must consent to provide data for the registry and must be willing to be contacted/reminded about data entry at each follow-up time point.
* Healthcare workers must agree to provide a secondary contact for follow-up.

Exclusion Criteria:

* A confirmed SARS-CoV-2 infection or clinically diagnosed COVID-19 prior to the first known exposure to confirmed or clinically diagnosed COVID-19 patient (Index Date).
* Participation in a 'blinded' clinical trial, i.e. unaware of exact treatment received as part of the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: As per the WHO definition10, HCWs eligible for enrollment are limited, based on the high likelihood of being exposed to COVID-19 patients during patient care, to the following positions:
  * Medical doctors*
  * Clinical officers*
  * Licensed physician assistant or nurse practitioner*
  * Registered nurse (or equivalent)*
  * Assistant nurse, nurse technician (or equivalent)*
  * Phlebotomist
  * Clinical pharmacist
  * Clinical physical therapist
  * Respiratory therapist
  * Community healthcare worker
    *These should include the following primary specialties:
  * Surgery (all sub-specialties)
  * Internal medicine (general)
  * Pulmonology/critical care
  * Emergency medicine
  * Geriatrics
  * Cardiology
  * Infectious disease
  * Anesthesiology
  * Pediatrics
  * Obstetrics/Midwifery
  * Other
Sampling Method: Non-Probability Sample
Enrollment: 6808 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Occurrence of SARS-CoV-2 infection among HCWs caring for COVID-19 patients, in terms of time, geography, healthcare setting, type of HCW. | 12 weeks
  Assess the association of potential prophylactic treatments with reduced risk of COVID-19 (or SARS-CoV-2 infection) in HCWs caring for COVID-19 patients

SECONDARY OUTCOMES:
Occurrence of SARS-CoV-2 uninfected HCWs | 12 weeks
  Subjects reporting "No" clinical diagnosis of COVID-19 or positive test results.
Occurrence of SARS-CoV-2 infection with ambulatory status and no limitation of activities | 12 weeks
  Subjects reporting COVID-19 related symptoms, clinical diagnosis of COVID-19 or positive test results but reporting "No" limitation of activities due to their symptoms and no hospitalization.
Occurrence of SARS-CoV-2 infection with ambulatory status and limitation of activities | 12 weeks
  Subjects reporting COVID-19 symptoms, clinical diagnosis of COVID-19 or positive test results and reporting "Yes" to having their usual activities limited being limited due to their symptoms, but no hospitalization.
Occurrence of hospitalization due to COVID-19 illness with mild disease | 12 weeks
  Subjects being hospitalised without being admitted to the ICU or without ventilation.
Occurrence of hospitalization due to COVID-19 illness with severe disease | 12 weeks
  Subjects being hospitalised with either admittance to the ICU and/or receiving ventilation.
Occurrence of all-cause mortality | 12 weeks
  Assess occurrence of all-cause mortality.
Type of prophylactic treatments by dose, frequency and duration, overall and by country/region/site | 12 weeks
  Assess the association between prophylactic treatments and the risk of SARS-CoV-2 infection in HCWs caring for COVID-19 patients.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Casciano, Masters, Principal Investigator — Certara; Craig Rayner, PharmD, Principal Investigator — Certara
Locations (1):
- Aga Khan University, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Providing survey response mapping, serology results, and technical report on an open access platform (Vivli)
Supporting Information: Study Protocol, SAP
Time Frame: Available on the Vivli - Center for Global Clinical Research platform
Access Criteria: Open access
URL: https://vivli.org/

DOCUMENTS (2):
  • Study Protocol (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT04626076/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-26): https://cdn.clinicaltrials.gov/large-docs/76/NCT04626076/SAP_001.pdf